CLINICAL TRIAL: NCT02448914
Title: A Single Centre, Two-period, Open Label, Randomised, Cross-over Study to Assess Plasma Levodopa, Carbidopa and Entacapone Concentrations After Continuous Infusion of TRIGEL or Duodopa in Patients With Advanced Parkinson´s Disease
Brief Title: A Study to Compare Plasma Levels of Levodopa, Carbidopa and Entacapone After TRIGEL or Duodopa Infusion in PD Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LobSor Pharmaceuticals AB (Industry)
Collaborators: TFS Trial Form Support (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: LSM-003; 2014-004891-46 (EudraCT Number)
Record Dates: First submitted 2015-05-12; First posted 2015-05-20 (Estimated); Results first posted 2016-05-23 (Estimated); Last update posted 2016-05-23 (Estimated); Status verified 2016-04

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — carbidopa, levodopa drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TRIGEL first, then Duodopa (Experimental): First Intervention (Day 1): TRIGEL, intestinal gel (20 mg/mL levodopa, 5 mg/mL carbidopa monohydrate, and 20 mg/mL entacapone).
  Second Intervention (Day 2): Duodopa, intestinal gel (20 mg/mL levodopa and 5 mg/mL carbidopa monohydrate).
  Both TRIGEL and Duodopa treatment consists of 3 individually adjusted and pre-defined doses: a morning dose, a continuous 14 h infusion, and extra bolus doses (if required).
  All TRIGEL doses correspond to 80% of the pre-study individually optimised doses of Duodopa. All Duodopa doses correspond to 100% of the pre-study individually optimized doses of Duodopa.
  Administration is done through duodenal or upper jejunal infusion via the patient's permanently inserted gastrojejunostomy tube by means of an ambulatory infusion pump.
  Interventions: Drug: TRIGEL; Drug: Duodopa
- Duodopa first, then TRIGEL (Experimental): First Intervention (Day 1): Duodopa, intestinal gel (20 mg/mL levodopa and 5 mg/mL carbidopa monohydrate).
  Second Intervention (Day 2): TRIGEL, intestinal gel (20 mg/mL levodopa, 5 mg/mL carbidopa monohydrate, and 20 mg/mL entacapone).
  Both TRIGEL and Duodopa treatment consists of 3 individually adjusted and pre-defined doses: a morning dose, a continuous 14 h infusion, and extra bolus doses (if required).
  All TRIGEL doses correspond to 80% of the pre-study individually optimised doses of Duodopa. All Duodopa doses correspond to 100% of the pre-study individually optimized doses of Duodopa.
  Administration is done through duodenal or upper jejunal infusion via the patient's permanently inserted gastrojejunostomy tube by means of an ambulatory infusion pump.
  Interventions: Drug: TRIGEL; Drug: Duodopa

INTERVENTIONS:
Drug: TRIGEL — All patients will receive TRIGEL. Treatment order is determined by randomization.
  Other Names: Lecigon
Drug: Duodopa — All patients will receive Duodopa. Treatment order is determined by randomization.
  Other Names: Duopa

SUMMARY:
This study evaluates the continuous addition of entacapone to infused levodopa and carbidopa on the pharmacokinetic (PK) profile in patients with advanced Parkinson's disease (PD). All patients will receive both study drugs, i.e. TRIGEL (levodopa, carbidopa, and entacapone) and Duodopa (levodopa and carbidopa), in randomized order.

DETAILED DESCRIPTION:
Intestinal infusion of Duodopa (levodopa and carbidopa) provides faster absorption, comparable levodopa bioavailability and significantly reduced intra-patient variability in levodopa concentrations relative to oral administration. TRIGEL also contains a third ingredient, entacapone. In tablet form, entacapone is shown to improve the bioavailability of levodopa and might extend the half-life of levodopa, avoiding deep troughs in levodopa plasma levels, and providing more continuous delivery of levodopa to the brain.

The intention with the study is to confirm that TRIGEL administration increases the area under the curve (AUC) for levodopa by combining levodopa, carbidopa, and entacapone and thereby lower the daily levodopa dose needed. It is expected that TRIGEL administration will result in a similar intra-patient variability in plasma levodopa concentrations as Duodopa during continuous administration.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide informed consent and judged by the Investigator to have decision-making capacity
2. Advanced levodopa-responsive idiopathic PD currently treated with Duodopa infusion since minimum 30 days
3. 30 years of age or older
4. BMI between 17.0 and 31.0 kg/m2, both inclusive
5. Agreed to use adequate contraceptive measures:

Female patients who have been post-menopausal for more than one year or female patients of childbearing potential using a highly efficient method of contraception during the study (i.e. a method with less than 1% failure rate [e.g. sterilisation, hormone implants, hormone injections, some intrauterine devices, or vasectomised partner]). Oral contraceptives in combination with other contraceptives are accepted.

Male patients being vasectomised or agreeing to use condoms during the study and having a partner who is using a highly efficient method of contraception as described above.

Exclusion Criteria:

1. Hypersensitivity or allergy to the investigational medicinal product (IMP) or to chemically related products
2. Contraindications for the use of levodopa or carbidopa or entacapone
3. Needing a daily total dose of Duodopa during study participation exceeding 125 mL
4. Increased fluctuation in clinical PD symptoms within 7 days prior to Screening
5. Administration of an investigational drug within 3 months prior to Screening and/or current participation in another clinical study involving a pharmaceutical or a medical device class III
6. Use of any forbidden medication as specified in Section 9.6 of the protocol
7. Known hepatitis B, hepatitis C or HIV infection
8. Donation of blood or plasma or major blood loss (≥500 mL) within 3 months prior to Screening
9. Positive urine drug test (amphetamine, benzodiazepines, tetrahydrocannabinol, cocaine or opiates) at Screening
10. Known alcohol abuse
11. Unwilling to meet the requirements of the protocol
12. Other medical or social reasons for exclusion at the discretion of the Investigator

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2015-05; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dag Nyholm, Assoc. Prof., Principal Investigator — Department of Neuroscience, Neurology, Uppsala University Hospital, Sweden
Locations (1):
- Clinical Trial Consultants AB, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- TRIGEL First, Then Duodopa: First Intervention (Day 1): TRIGEL, intestinal gel (20 mg/mL levodopa, 5 mg/mL carbidopa monohydrate, and 20 mg/mL entacapone).
  Second Intervention (Day 2): Duodopa, intestinal gel (20 mg/mL levodopa and 5 mg/mL carbidopa monohydrate).
  Both TRIGEL and Duodopa were administered during 14 h in total. Each treatment consisted of three individually adjusted and pre-defined doses: a morning dose, a continuous administration, and extra doses (if required).
  The TRIGEL doses corresponded to 80% of the pre-study individually optimized doses of Duodopa in the first cohort of 5 patients. After the first cohort, a pre-planned interim analysis was performed. It was decided that the morning dose would be adjusted from 80% to 90% of the corresponding Duodopa dose for the second cohort. No other changes to the dosage regimens were made. All Duodopa doses corresponded to 100% of the pre-study individually optimized doses of Duodopa.
- Duodopa First, Then TRIGEL: First Intervention (Day 1): Duodopa, intestinal gel (20 mg/mL levodopa and 5 mg/mL carbidopa monohydrate).
  Second Intervention (Day 2): TRIGEL, intestinal gel (20 mg/mL levodopa, 5 mg/mL carbidopa monohydrate, and 20 mg/mL entacapone).
  Both TRIGEL and Duodopa were administered during 14 h in total. Each treatment consisted of three individually adjusted and pre-defined doses: a morning dose, a continuous administration, and extra doses (if required).
  The TRIGEL doses corresponded to 80% of the pre-study individually optimized doses of Duodopa in the first cohort of 5 patients. After the first cohort, a pre-planned interim analysis was performed. It was decided that the morning dose would be adjusted from 80% to 90% of the corresponding Duodopa dose for the second cohort. No other changes to the dosage regimens were made. All Duodopa doses corresponded to 100% of the pre-study individually optimized doses of Duodopa.
Period: First Intervention (1 Day)
Arm/Group | TRIGEL First, Then Duodopa | Duodopa First, Then TRIGEL
Started | 6 | 5
Completed | 6 | 5
Not Completed | 0 | 0
Period: Second Intervention (1 Day)
Arm/Group | TRIGEL First, Then Duodopa | Duodopa First, Then TRIGEL
Started | 6 | 5
Completed | 6 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- TRIGEL and Duodopa in Randomized Order: TRIGEL, intestinal gel (20 mg/mL levodopa, 5 mg/mL carbidopa monohydrate, and 20 mg/mL entacapone). Duodopa, intestinal gel (20 mg/mL levodopa and 5 mg/mL carbidopa monohydrate).
  All patients received TRIGEL and Duodopa treatment on two consecutive days in the study. Both TRIGEL and Duodopa were administered during 14 h in total. Each treatment consisted of three individually adjusted and pre-defined doses: a morning dose, a continuous administration, and extra doses (if required).
  The TRIGEL doses corresponded to 80% of the pre-study individually optimized doses of Duodopa in the first cohort of 5 patients. After the first cohort, a pre-planned interim analysis was performed. It was decided that the morning dose would be adjusted from 80% to 90% of the corresponding Duodopa dose for the second cohort. No other changes to the dosage regimens were made. All Duodopa doses corresponded to 100% of the pre-study individually optimized doses of Duodopa.
Arm/Group | TRIGEL and Duodopa in Randomized Order
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 10
Age, Continuous [Mean (Full Range); unit: years] | 69.5 [63 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 7
Region of Enrollment [Number; unit: participants]
  Sweden | 11

OUTCOME MEASURES:

1. Primary Outcome: Dose Adjusted Area Under the Curve (AUC) (0-14h) for Levodopa
Time Frame: During 14 h infusion on 2 consecutive days
Measure: Least Squares Mean (Full Range); unit: h*ng/mL/mg
Groups:
- TRIGEL: TRIGEL, intestinal gel (20 mg/mL levodopa, 5 mg/mL carbidopa monohydrate, and 20 mg/mL entacapone).
  All patients received TRIGEL and Duodopa treatment on two consecutive days in the study.
  Both TRIGEL and Duodopa were administered during 14 h in total. Each treatment consisted of three individually adjusted and pre-defined doses: a morning dose, a continuous administration, and extra doses (if required).
  The TRIGEL doses corresponded to 80% of the pre-study individually optimized doses of Duodopa in the first cohort of 5 patients. After the first cohort, a pre-planned interim analysis was performed. It was decided that the morning dose would be adjusted from 80% to 90% of the corresponding Duodopa dose for the second cohort. No other changes to the dosage regimens were made.
- Duodopa: Duodopa, intestinal gel (20 mg/mL levodopa and 5 mg/mL carbidopa monohydrate).
  All patients received TRIGEL and Duodopa treatment on two consecutive days in the study. Both TRIGEL and Duodopa were administered during 14 h in total. Each treatment consisted of three individually adjusted and pre-defined doses: a morning dose, a continuous administration, and extra doses (if required).
  All Duodopa doses corresponded to 100% of the pre-study individually optimized doses of Duodopa.
Arm/Group | TRIGEL | Duodopa
Number analyzed (Participants) | 11 | 11
h*ng/mL/mg | 40.6 [22.3 to 69.4] | 29.4 [21.7 to 52.8]
Statistical Analysis 1: Comparison: TRIGEL vs Duodopa; Levodopa AUC 0-14h/dose, was derived using the trapezoidal method and divided by the total administered dose of levodopa during the corresponding time interval.The primary endpoint was log transformed and analysed using an ANCOVA, adjusting for treatment, period and patient. The back-transformed ratio of TRIGEL over Duodopa was calculated together with 95% confidence intervals (CI) and the associated (2 sided) p value; Test type: Non-Inferiority or Equivalence — Analysis was first to attempt to show non-inferiority. To show non-inferiority of TRIGEL over Duodopa, the lower limit of the two-sided CI for the treatment ratio had to be above the chosen non-inferiority margin of 0.9. If non-inferiority was shown, analysis continued with test of superiority. To show superiority of TRIGEL versus Duodopa, the lower confidence limit had to be above 1 (corresponding to a p-value less than 0.05); p < 0.0001, ANCOVA; back-transformed ratio = 1.382, 95% CI 2-sided [1.264 to 1.511]

2. Secondary Outcome: Intra-individual Coefficient of Variation (3-14h) for Levodopa
Description: The individual patient's coefficient of variation (CV) of levodopa plasma concentration during administration of TRIGEL and Duodopa respectively between 3 and 14 h after start of study drug. CV=100*sqrt (exp (SDlog*SDlog)-1) were SDlog denotes the standard deviation computed on logged plasma concentrations.
Time Frame: During 3-14h infusion on 2 consecutive days
Measure: Least Squares Mean (Full Range); unit: percentage of variability
Arm/Group | TRIGEL | Duodopa
Number analyzed (Participants) | 11 | 11
percentage of variability | 13.8 [6.5 to 36.7] | 10.6 [6.1 to 19.2]

3. Secondary Outcome: Dose Adjusted AUC (0-14h) for Carbidopa
Time Frame: During 14 h infusion on 2 consecutive days
Measure: Least Squares Mean (Full Range); unit: h*ng/mL/mg
Arm/Group | TRIGEL | Duodopa
Number analyzed (Participants) | 11 | 11
h*ng/mL/mg | 22.1 [13.6 to 52.5] | 18.8 [11.5 to 37.9]

4. Secondary Outcome: Number of Adverse Events
Time Frame: Patients will be followed for the duration of the hospital stay, an expected average of 3 days
Measure: Number; unit: adverse events
Arm/Group | TRIGEL | Duodopa
Number analyzed (Participants) | 11 | 11
adverse events | 10 | 6

5. Secondary Outcome: Dose Adjusted AUC (0-14h) for 3-O-Methyldopa
Time Frame: During 14 h infusion on 2 consecutive days
Measure: Least Squares Mean (Full Range); unit: h*ng/mL/mg
Arm/Group | TRIGEL | Duodopa
Number analyzed (Participants) | 11 | 11
h*ng/mL/mg | 155 [83.9 to 258.3] | 131 [72.1 to 182.2]

6. Other Pre Specified Outcome: Treatment Response Scale (ON/OFF Effect) - Mean % of Time Patients Were in Functional ON State During 3-14 h
Description: Dyskinesia and parkinsonism symptoms were evaluated throughout the study period as an assessment of the clinical response. To assess the ON/OFF effect the Treatment Response Scale (TRS) was used. The TRS ranges from -3 (severe "OFF") to +3 ("ON" with severe dyskinesia). Results from the TRS recordings are presented as the mean percentage of time patients were in functional ON state (TRS: -1 to +1) during the time interval 3-14 h.
Time Frame: TRS assessments were made every 30 minutes from start of study drug administration until 3 h, every hour between 3 and 14 h and every 30 minutes between 14 and 17 h.
Measure: Mean (Full Range); unit: Mean % of time
Arm/Group | TRIGEL | Duodopa
Number analyzed (Participants) | 11 | 11
Mean % of time | 91.7 [18.3 to 100.0] | 91.0 [0.758 to 100.0]

ADVERSE EVENTS:
Arm/Group | TRIGEL | Duodopa
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 6/11 | 2/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TRIGEL (N=11) | Duodopa (N=11)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (2)
Injection site haematoma (Injury, poisoning and procedural complications) | 1 (3) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 1 (1)
Cold sweat (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other